CLINICAL TRIAL: NCT04122170
Title: A Phase 2B, Randomized, Double-blind, Multicenter, Placebo-controlled Study to Evaluate the Efficacy of Bentracimab (PB2452) in Reversing Ticagrelor in Subjects Aged 50 to 80 Years Old
Brief Title: Phase 2B Study to Evaluate the Efficacy of Bentracimab (PB2452) in Reversal of Ticagrelor in Subjects Aged 50-80 Years Old
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SFJ Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB2452-PT-CL-0003
Record Dates: First submitted 2019-10-04; First posted 2019-10-10 (Actual); Results first posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-02

CONDITIONS: Healthy
MeSH Terms: interventions — Aspirin; PB-2452; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bentracimab (PB2452) (Active Comparator): PB2452 18 g Intravenous Infusion over a 16 hour duration.
  Interventions: Drug: Ticagrelor Oral Tablet - Pre-Treatment; Drug: Aspirin (ASA) Oral Tablet - Pre-Treatment; Drug: Bentracimab (PB2452) Infusion
- Placebo (Placebo Comparator): Placebo (0.9% Sodium chloride) intravenous Infusion over a 16 hour duration.
  Interventions: Drug: Ticagrelor Oral Tablet - Pre-Treatment; Drug: Aspirin (ASA) Oral Tablet - Pre-Treatment; Drug: Placebo (0.9% Sodium chloride) infusion

INTERVENTIONS:
Drug: Ticagrelor Oral Tablet - Pre-Treatment — Ticagrelor 90 mg oral tablet; administered as 180 mg (2 × 90 mg tablet) loading dose plus 90 mg every 12 hours for 4 additional doses.
Drug: Aspirin (ASA) Oral Tablet - Pre-Treatment — Aspirin 81 mg oral tablet; administered daily between Day -7 to the morning before receiving study medication on Day 1, for a total of 8 tablets only.
Drug: Bentracimab (PB2452) Infusion — Bentracimab (PB2452) 18 g Intravenous Infusion over a 16 hour duration
  In subjects with potential drug interaction from concomitant use of moderate or strong CYP3A inhibitors with ticagrelor, the active treatment period may be 24 hours and 10 min if receiving the 36 g infusion.
  Arms: Bentracimab (PB2452)
Drug: Placebo (0.9% Sodium chloride) infusion — 0.9% Sodium chloride Intravenous Infusion over a 16 hour duration
  Arms: Placebo

SUMMARY:
This phase 2B study is a multi-center, randomized, double-blind, placebo-controlled study. The study is designed to evaluate the efficacy of bentracimab (PB2452) in reversing the anti-platelet effects of ticagrelor as part of a dual antiplatelet regimen and to evaluate the safety and tolerability of bentracimab (PB2452) in subjects aged 50-80 years old.

A total of 205 subjects between 50-80 years old will be enrolled in the US or other countries at the discretion of the Sponsor across 5-15 sites. The subjects will be randomized at a ratio of 3:1 receiving either the bentracimab (PB2452) investigational study drug or placebo. Hence, a total of 154 subjects will be receiving bentracimab (PB2452) and approximately 51 subjects will be receiving placebo.

DETAILED DESCRIPTION:
The study will consist of a Screening period, a Check-in day, an on-site Randomization/Treatment day, a 2-day on-site Follow-up period (Days 2 through 3), a Follow-up visit (Day 7), and a Final Follow-up visit (Day 35±3). If needed and at the discretion of the Investigator, a subject may remain in the study facility beyond the scheduled Day 3 discharge to accommodate Day 7 and Day 35±3 follow-up visits. Seven days prior to enrollment, subjects will be administered ASA 81 mg orally once daily (QD) until the final dose on Day 1. Beginning in the morning on Day -2, a single dose of oral ticagrelor 180 mg will be given, followed by oral ticagrelor 90 mg every 12 hours for 4 additional doses through to Day 1 (2 hours before study drug is initiated; this will be 5 total doses of ticagrelor).

On Day 1, subjects who meet all the inclusion criteria and none of the exclusion criteria will be randomized with 3:1 allocation ratio (active:placebo), to receive an IV dose of bentracimab (PB2452) or placebo 2 hours following the 5th ticagrelor dose. Subjects may be discharged from the clinical site on Day 3 and will return for a Follow-up visit on Day 7, if already discharged, and on Day 35 (±3 days). A subject may remain in the study facility beyond the scheduled Day 3 discharge to accommodate Day 7 and Day 35±3 follow-up visits.

If a subject is taking a moderate or strong cytochrome P450 3A isozyme (CYP3A) inhibitor, a 36 g alternative regimen of bentracimab (PB2452) will be administered consisting of 12 g infused over 10 minutes followed by a 12 g loading dose infused over 6 hours, then a maintenance dose of 12 g infused over the next 18 hours immediately following completion of the loading period for a total infusion time of approximately 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* The subject provides written or verbal informed consent (in-person or remotely) and agrees to comply with all protocol requirements throughout study participation.
* The subject is male or female between ≥50 and ≤80 years of age.
* The subject has a body mass index between 18 and 35 kg/m2 and a weight of ≥ 50 kg but ≤ 120 kg, inclusive, at screening.
* The subject is considered by the Investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12 lead ECG results, and physical examination findings at screening and Check-in. Subjects with chronic, stable, and well-controlled medical conditions, are eligible provided they meet all other inclusion/exclusion criteria.
* The subject has specific inclusionary laboratory values at screening and check-in: white blood cell (WBC) count, platelet count, haemoglobin level, thyroid-stimulating hormone (TSH) level, and prothrombin time (PT) and partial thromboplastin time (PTT) levels within the normal range.
* Subjects taking medications for well-controlled medical conditions must have been on a stable dose for at least 30 days prior to screening visit.
* Subjects entering the study must be willing to start and/or document an 81 mg daily dose of aspirin on Day -7 and must document daily dosing until the final dose is administered on the morning of Day 1. Subjects already taking daily aspirin must suspend aspirin dosing after Day 1 until discharge from the clinical facility.
* Female subjects of childbearing potential must not be pregnant, lactating, or planning to become pregnant for 3 months after the last dose of study drug. Female subjects of childbearing potential must use two effective methods of birth control from screening and before study drug administration through to the end of the study.

Exclusion Criteria:

* In the opinion of the Investigator there are concern(s) regarding the inability of the subject to comply with study procedures and/or follow up, or, if the subject is not suitable for entry into the study.
* History of any acute or chronic medical disorder expected to decrease the life expectancy of the subject to an extent where the subject's study participation is affected.
* Any clinically significant acute illness, medical/surgical procedure, or trauma within 4 weeks of the administration of study drug or any planned surgical procedure that will occur during the study.
* Any clinically significant abnormal findings in physical examination, vital signs, laboratory assessments, and ECG parameters identified during screening or check-in.
* Any specific contraindication to ticagrelor as described in the ticagrelor prescribing information.
* Receiving chronic treatment with nonsteroidal anti-inflammatory drugs [including aspirin (>100 mg daily), anticoagulants, or other antiplatelet agents that cannot be discontinued 14 days prior to screening including clopidogrel, prasugrel, ticlopidine, dipyridamole, or cilostazol].
* First positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies at screening.
* Has received another investigational drug within 30 days of the administration of study drug in this study or within 5 half-lives of the experimental medication, whichever is longer.
* History of severe or ongoing allergy/hypersensitivity to any biologic therapeutic agent.
* Involvement with any PhaseBio or study site employee or their close relatives (e.g., spouse, parents, siblings, or children whether biological or legally adopted).
* Previously received Bentracimab (PB2452) or had been randomized to receive study drug in an earlier cohort for this study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (13):
  - Woodland Research Northwest, LLC, Rogers, Arkansas
  - WCCT Global, Inc., Cypress, California
  - Pacific Research Network, San Diego, California
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - PPD Development, LP, Orlando, Florida
  - Altasciences Clinical Kansas, Inc., Overland Park, Kansas
  - BioPharma Services USA Inc. (BPSUSA), St Louis, Missouri
  - Monroe Biomedical Research, Monroe, North Carolina
  - Aventiv Research Inc., Columbus, Ohio
  - Remington-Davis, Inc., Columbus, Ohio
  - VitaLink Research - Greenville, Greenville, South Carolina
  - VitaLink Research - Spartanburg, Spartanburg, South Carolina
  - Rebecca Wood-Horrall, Austin, Texas
- Canada (2):
  - BioPharma Services Inc., Toronto, Ontario
  - Altasciences Company Inc., Mount Royal, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bentracimab (PB2452): PB2452 18 g Intravenous Infusion over a 16 hour duration.
  Ticagrelor Oral Tablet - Pre-Treatment: Ticagrelor 90 mg oral tablet; administered as 180 mg (2 × 90 mg tablet) loading dose plus 90 mg every 12 hours for 4 additional doses.
  Aspirin (ASA) Oral Tablet - Pre-Treatment: Aspirin 81 mg oral tablet; administered daily between Day -7 to the morning before receiving study medication on Day 1, for a total of 8 tablets only.
  Bentracimab (PB2452) Infusion: Bentracimab (PB2452) 18 g Intravenous Infusion over a 16 hour duration
  In subjects with potential drug interaction from concomitant use of moderate or strong cytochrome P450 3A isozyme (CYP3A) inhibitors with ticagrelor, the active treatment period may be 24 hours and 10 min if receiving the 36 g infusion.
Period: Overall Study
Arm/Group | Bentracimab (PB2452) | Placebo
Started | 156 | 51
Completed | 150 | 50
Not Completed | 6 | 1

BASELINE CHARACTERISTICS:
Population: There were initially 207 subjects randomized but 2 of these subjects were randomized in error and did not receive study drug.
Groups:
- Bentracimab (PB2452): PB2452 18 g Intravenous Infusion over a 16 hour duration.
  Ticagrelor Oral Tablet - Pre-Treatment: Ticagrelor 90 mg oral tablet; administered as 180 mg (2 × 90 mg tablet) loading dose plus 90 mg every 12 hours for 4 additional doses.
  Aspirin (ASA) Oral Tablet - Pre-Treatment: Aspirin 81 mg oral tablet; administered daily between Day -7 to the morning before receiving study medication on Day 1, for a total of 8 tablets only.
  Bentracimab (PB2452) Infusion: Bentracimab (PB2452) 18 g Intravenous Infusion over a 16 hour duration
  In subjects with potential drug interaction from concomitant use of moderate or strong CYP3A inhibitors with ticagrelor, the active treatment period may be 24 hours and 10 min if receiving the 36 g infusion.
- Total: Total of all reporting groups
Arm/Group | Bentracimab (PB2452) | Placebo | Total
Number analyzed (Participants) | 154 | 51 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (6.90) | 60.9 (6.76) | 61.2 (6.85)
Age, Customized [Count of Participants; unit: Participants]
  <= 65 years | 107 | 39 | 146
  > 65 years | 47 | 12 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 30 | 102
  Male | 82 | 21 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 7 | 25
  Not Hispanic or Latino | 136 | 44 | 180
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 8 | 37
  White | 121 | 43 | 164
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 23 | 8 | 31
  United States | 131 | 43 | 174
Renal Group [Count of Participants; unit: Participants] — Population: Number of subjects with observation at baseline.
  Participants
    number analyzed (Participants) | 151 | 50 | 201
    Normal | 46 | 16 | 62
    Mild | 91 | 30 | 121
    Moderate | 14 | 4 | 18
    Severe | 0 | 0 | 0
    ESRD | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: Kilograms] | 80.8 (14.77) | 80.4 (12.93) | 80.7 (14.30)
Height [Mean (Standard Deviation); unit: Centimeters] | 169.9 (10.17) | 168.3 (9.99) | 169.5 (10.12)
BMI [Mean (Standard Deviation); unit: kilograms/meters^2] | 27.9 (3.71) | 28.3 (3.49) | 28.0 (3.65)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Minimum Percent Inhibition Platelet Reactivity Unit (PRU) Assessed by VerifyNow™ PRUTest™ From Baseline to Within 4 Hours After Study Drug Start.
Description: Reversal of anti-platelet effects of ticagrelor with intravenous infusion of bentracimab (PB2452) or placebo
Time Frame: Baseline (pre-dose) to 4 hours after the start of infusion
Measure: Mean (95% Confidence Interval); unit: Percent Inhibition of PRU Over 4 Hours
Arm/Group | Bentracimab (PB2452) | Placebo
Number analyzed (Participants) | 154 | 51
Percent Inhibition of PRU Over 4 Hours | -5.99 [-8.55 to -3.43] | 90.11 [86.24 to 93.98]

ADVERSE EVENTS:
Time Frame: Through End of Study Visit (Day 35)
Description: Serious Adverse Events (SAEs) and Adverse Events (AEs) reported for Safety Subset which includes subjects who received any amount of study drug; 2 subjects randomized in error and did not receive study drug. Subjects could spontaneously report and/or were asked a standard question to elicit any medically related changes in well-being. Changes in lab values, physical exam findings, 12-lead ECG monitoring changes, or other events relevant to subject safety were assessed and reported as an AE.
Arm/Group | Bentracimab (PB2452) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/156 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/154 | 1/51
Other Adverse Events (participants affected / at risk) | 58/154 | 21/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bentracimab (PB2452) (N=154) | Placebo (N=51)
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bentracimab (PB2452) (N=154) | Placebo (N=51)
Vessel puncture site bruise (General disorders) | 4 | 1
Oedema (General disorders) | 2 | 1
Catheter site bruise (General disorders) | 1 | 1
Infusion site extravasation (General disorders) | 2 | 0
Administration site bruise (General disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 1 | 0
Catheter site oedema (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Crepitations (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Infusion site bruising (General disorders) | 0 | 1
Infusion site erythema (General disorders) | 1 | 0
Infusion site pruritus (General disorders) | 1 | 0
Infusion site reaction (General disorders) | 0 | 1
Injection site haemorrhage (General disorders) | 1 | 0
Injection site phlebitis (General disorders) | 1 | 0
Injection site reaction (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Thirst (General disorders) | 0 | 1
Vessel puncture site erythema (General disorders) | 1 | 0
Headache (Nervous system disorders) | 6 | 4
Dizziness (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 2
Oral disorder (Gastrointestinal disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 5 | 2
Burns first degree (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 6 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Occult blood (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Occult blood positive (Investigations) | 1 | 0
Asymptomatic COVID-19 (Infections and infestations) | 2 | 0
COVID-19 (Infections and infestations) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT04122170/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT04122170/SAP_001.pdf